CLINICAL TRIAL: NCT04140760
Title: Can a 12-week Probiotic Intervention Improve Wellbeing in Parkinson's Disease? A Randomised Double-blind Placebo-controlled Feasibility Study
Brief Title: Probiotic Use in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sheffield Hallam University (Other)
Collaborators: University of Sheffield (Other); Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 262286
Record Dates: First submitted 2019-09-20; First posted 2019-10-28 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Study is double blind design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Active Comparator): Thirty five Parkinson's Disease patients group will be randomly assigned to this study arm.
  Participants will take the liquid probiotic (Symprove) daily following manufacturers guidelines for a period of 12 weeks.
  Interventions: Other: Symprove
- Placebo (Placebo Comparator): Thirty five Parkinson's Disease patients group will be randomly assigned to this study arm.
  Participants will take the liquid placebo daily for a period of 12 weeks following the same guidelines as for the probiotic.
  Interventions: Other: Symprove placebo product

INTERVENTIONS:
Other: Symprove — A liquid probiotic
  Arms: Probiotic
Other: Symprove placebo product — An inert placebo
  Arms: Placebo

SUMMARY:
1. To evaluate the components and processes needed for a full-scale clinical study: recruitment, randomisation, attrition, probiotic use, stool sample collection, microbiome sequencing and behavioural/cognitive measures and determine the feasibility and patient acceptability of these processes to inform a full-scale study in line with NIHR pilot study guidance.
2. To collect pilot data to determine sample size and power, reliability and sensitivity of selected measures, to maximise the findings and minimise patient burden.

DETAILED DESCRIPTION:
The proposed research is a pilot study with 70 participants, 35 in the probiotic and 35 in the placebo arm of the study. The study will investigate the process of conducting randomised, double-blind, placebo-controlled research about probiotic use in Parkinson's Disease patients. The primary aim of the study is to test elements of the study design for a full-scale clinical study: recruitment, randomisation, probiotic use, stool sample collection and DNA sequencing and behavioural/cognitive measures. The secondary aim is to collect pilot data to determine the sample size, Power and appropriateness of measures needed for a full-scale study that maximises findings and minimises patient burden.

Parkinson's Disease (PD) is a neurodegenerative condition that affects motor functions and a range of non-motor abilities. There is no cure and a definitive cause is not yet known. It has a prevalence of 0.3% in the general population and 1-3% in the population over the age of 65. Globally, it is the second most common neurodegenerative disorder and due to the lack of early diagnosis and effective therapy, represents a large burden for society and healthcare provision. The underlying pathology of PD is associated with accumulation of abnormal clumps of alpha-synuclein protein termed Lewy bodies and Lewy neurites in the central nervous system (CNS) that impede the normal function of brain cells. Evidence from animal studies indicates that the production of alpha-synuclein begins in the gut, and gastro-intestinal problems are a common feature of PD.

The gut contains millions of micro-organisms termed the microbiome. Over the past decade research findings have identified a complex bidirectional interaction between the gastrointestinal (GI) tract and the central nervous system (CNS), the Gut-Brain axis. It is now known that the Gut-Brain axis is adversely affected by PD. Recently, probiotics have been proposed as a potential intervention for systemic and neurological conditions by improving microbiome composition.

Data obtained from this pilot study will be used to identify challenges in conducting research using probiotics in patients with Parkinson's Disease and provide a rationale for conducting a full-scale study including information that may reduce or eliminate problems that limit the successful delivery of a full-scale trial. The investigators will make no claims here about any purported clinical effects of the chosen probiotic.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's disease based on UK PD Society Brain Bank criteria.
* Capacity to consent and complete questionnaires.
* Absence of gut/intestinal disorders that would prevent use of a probiotic and/or cause diarrhoea.
* Absence of coincidental neurological condition.
* Using l-dopa plus or minus a dopaminergic agonist.
* Age over 18 and under 80

Exclusion Criteria:

* Unable to consent.
* Use of systemic antibiotics, antifungals, antivirals or antiparasitics (intravenous, intramuscular, or oral).
* Use of commercial probiotics: includes tablets, capsules, lozenges, chewing gum or powders in which probiotic is a primary component. Ordinary dietary components such as fermented beverages/milks, yogurts, foods do not apply.
* Presence of acute viral/bacterial infection disease at the time of sampling (defer sampling until subject recovers). Acute disease is defined as the presence of a moderate or severe illness with or without fever.
* Major surgery of the GI tract, with the exception of cholecystectomy and appendectomy, in the past five years. Any major bowel resection at any time.
* History of active uncontrolled gastrointestinal disorders or diseases including: inflammatory bowel disease (IBD) including ulcerative colitis (mild-moderate-severe), Crohn's disease (mild-moderate-severe), or indeterminate colitis.
* Presence of persistent, infectious gastroenteritis, colitis or gastritis, persistent or chronic diarrhea of unknown etiology, Clostridium difficile infection (recurrent) or Helicobacter pylori infection (untreated).
* Presence of incidental neurological illness.
* Experience of any type of cancer or adenoma less than 5 years previously.
* Age over 80

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-08-14 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-12-22 (Estimated)

PRIMARY OUTCOMES:
Patient Adherence to Study questionnaire | Thirteen weeks from study start
  The patient experience questionnaire (Adherence To Study) provides data about patients' experience of taking part in the study to inform a full-scale trial. These data will enable evaluation of the patient experience of taking part in the study, the experience of providing two stool samples and taking a daily capful of the placebo or probiotic liquid. This scale is developed by the researcher's. The measure is a 5-point Likert scale that includes responses: Not at all, 2 = Not really, 3 = Somewhat, 4 = Quite a lot, 5 = Very much - in the first part of the questionnaire. A sample question is: Are you happy with the consent process for taking part in the research? Total score ranges from 6-30 - low score indicates dissatisfaction with the study method and information provided. Other questions in the scale require simple 'yes' and 'no' responses. For example, 'Were you comfortable providing a stool sample for the study?'
Patient Exit Study Scale | 12 and 24 weeks from study start date (only relevant for patients who withdrew).
  The patient exit study scale is designed to evaluate why patients did not or were unable to complete the study. The scale was devised by the researchers and comprised a 5-point Likert scale. Scores range from 7-35 with lower scores indicating dissatisfaction with particular elements of of study design, recruitment, and/or data collection. These data will inform the full-scale study

SECONDARY OUTCOMES:
Microbiome measurement: 16S rRNA gene sequencing and compositional analysis Microbiome measurement: 16S rRNA gene sequencing and compositional analysis for each patient at pre- and post-intervention | First sample taken at week 1 of entry into study; second sample taken at week 13 after entry to study.
  A total of 140 samples for16S rRNAv4 Gene Sequencing and analysis n = 35 in each group, two groups (baseline and after probiotics/placebo treatment). Each patient will have two samples collected before and after probiotics/placebo treatment. Stool samples will be shipped to Diversigen (USA) for DNA extraction and sequencing
The Unified Parkinson's disease rating scale (UPDRS): Fahn S, Elton R, UPDRS 1987, pp 153-163, 293-304 | Measure to be completed at week 1 of entry into study; second evaluation completed at week 13 after entry to study.
  The UPDRS workbook measures: I. Mentation, Behaviour, Mood - Four Subscales: Range 0-4 Total range = 0-16. II. Activities of daily living - Thirteen Subscales: Range 0-4 Total: 0-52. III. Motor Examination - Fourteen Subscales: Range 0-4 Total range 0-56. Zero = absence of symptoms, 4 = most severe presence of symptoms for all scales. Hoehn and Yahr Staging scale 0-5 (0 = no symptoms, 5 = wheelchair bound or bedridden.
The Parkinson's Disease Questionnaire (PDQ-39) Quality of Life Scale | Measure to be completed at week 1 of entry into study; second evaluation completed at week 13 after entry to study.
  The user manual specifies that the questionnaire is particularly appropriate for use in clinical trials to assess treatments and interventions intended to benefit people with Parkinson's disease. Scale is 5-point Likert scale from 'Never' through to 'Always' with scores ranging from 0-4. Total score range = 0 - 156 (Lower score = better quality of life, higher score = poorer quality of life.
The Parkinson's Disease Sleep Scale | Measure to be completed at week 1 of entry into study; second evaluation completed at week 13 after entry to study.
  The PDSS is a visual analogue scale addressing 15 commonly reported symptoms associated with sleep disturbance. Response options range from 0 = 'awful' to 10 = 'excellent' or 0 = 'always' to 10 = 'never.' Total score range from 0-150. Low scores indicate poor sleep or sleep related problems and high scores indicate good sleep quality.
Gastrointestinal Symptom Rating Scale (GSRS) | Measure to be completed at week 1 of entry into study; second evaluation completed at week 13 after entry to study.
  This measure includes questions relating to 15 common gastrointestinal symptoms and requires patients to rate the severity of their symptoms over the past week or 2 weeks. It was developed from reviews of gastrointestinal symptoms and clinical experience, to evaluate common symptoms of gastrointestinal disorders. Responses range from 1 = 'No discomfort at all' to 7 = 'Very severe discomfort.' Total score range is 15-105, where 15 indicates minimal discomfort and higher rating scores indicate significant or severe discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Lynne A Barker, BSc (hons) PhD, Principal Investigator — Sheffield Hallam University
Locations (1):
- Sheffield Hallamshire Hospital, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No